CLINICAL TRIAL: NCT03654937
Title: Immune Response and Risk of Side Effects After Influenza Vaccination in Athletes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universität des Saarlandes (Other)
Collaborators: Federal Institute of Sport Science (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Impftrain
Record Dates: First submitted 2018-08-30; First posted 2018-08-31 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Influenza Virus Vaccine Adverse Reaction; Influenza Vaccine Allergy
Keywords: Influenza vaccination; elite athletes; Immune response; Side effects
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 2h (Active Comparator): The participants were asked to report for their vaccination immediately after an intensive bout of training (not later than two hours after). The influenza vaccine was administered via intra-muscular injection into the deltoid muscle of the non-dominant arm in a standardized manner.
  Interventions: Biological: Influenza Vaccination
- 26h (Active Comparator): The athletes of the second group were vaccinated after an entire day (between 24 and 26 hours) after their last training session.The vaccine was administered via intra-muscular injection into the deltoid muscle of the non-dominant arm in a standardized manner.
  Interventions: Biological: Influenza Vaccination

INTERVENTIONS:
Biological: Influenza Vaccination — Influenza vaccination "Influsplit Tetra" 2016/2017, GlaxoSmithKline GmbH & Co. KG, Munich, Germany, batch: AFLBA 152AB.

SUMMARY:
Seasonal influenza vaccination was used to assess whether induction of immunity as well as the rate of side effects is influenced by the timing of the last training session before vaccination. Healthy athletes were vaccinated with the tetravalent influenza vaccine and blood samples were collected before, 1, 2 and 26 weeks after vaccination. The athletes were randomly assigned to vaccination within 2 hours after the last training session ("2h") vs. vaccination after a resting period of at least 26 hours ("26h"). All participants documented side effects and training restrictions. Influenza-specific T-cells were quantified after stimulation with the vaccine based on intracellular cytokine staining. Antibodies were quantified by ELISA and neutralisation assay.

ELIGIBILITY:
Inclusion Criteria:

* performance-oriented training on at least five days a week, healthy athletes

Exclusion Criteria:

* current acute infection, allergy to the vaccine, immunosuppression, pregnancy, rheumatic diseases

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2018-04-01 (Actual)

PRIMARY OUTCOMES:
Immune response | 26 weeks
  Influenza-specific T-cells were quantified after stimulation with the vaccine based on intracellular cytokine staining. Antibodies were quantified by ELISA and neutralisation assay.
Rate of side effects | 2 weeks
  All participants documented side effects and training restrictions.